CLINICAL TRIAL: NCT06565221
Title: Microvascular Blood Flow During Passive Heating
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-2024-0167
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Blood Flow

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat and negative pressure (Experimental): Forearm and quadriceps blood flow at baseline and during intervention
  Interventions: Device: Heat and negative pressure

INTERVENTIONS:
Device: Heat and negative pressure — Heat and negative pressure applied to the feet

SUMMARY:
Determine whether passive heating intervention effects microvascular blood flow as measured with near-infrared spectroscopy

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 50 years

Exclusion Criteria:

* Diagnosis of peripheral neuropathy
* open wounds on feet

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Microvascular blood flow volume | Baseline and during intervention
  Measured using NIRS